CLINICAL TRIAL: NCT03208855
Title: Cognitive Behavioral Therapy for Insomnia in Substance Use Disorders at an Urban Residential Recovery Program
Brief Title: Cognitive Behavioral Therapy for Insomnia in Substance Use Disorders
Acronym: gCBTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00117179
Record Dates: First submitted 2017-06-28; First posted 2017-07-06 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Substance Use Disorders; Insomnia
Keywords: Cognitive Behavioral Therapy
MeSH Terms: conditions — Substance-Related Disorders; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I (Experimental): Participants will receive 8 1-hour sessions of group Cognitive Behavioral Therapy for insomnia as part of their intensive outpatient treatment of substance use recovery
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
- Treatment as Usual (No Intervention): Participants will receive treatment as usual for substance abuse treatment as part of their intensive outpatient treatment of substance use recovery

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — 8 week 1-hour sessions of group CBT-I with each group including 3-4 men.
  Other Names: gCBT-I
  Arms: CBT-I

SUMMARY:
Substance Use Disorders (SUDs) and insomnia are major public health concerns, and each are independently linked to reduced quality of life, disability, and high healthcare costs. Insomnia, characterized by difficulty initiating or maintaining sleep, or nonrestorative sleep, is prevalent in 10% of the general population and is co-morbid in 70% of patients with SUDs. Primary insomnia and SUDs are chronic, unremitting diseases and have a complex bidirectional relationship. Insomnia symptoms may predate the onset of SUDs and may explain high prevalence of self-treatment. Insomnia may also be a direct effect of intoxication, withdrawal, or abstinence from the substance of abuse. Subjective and objective measures of sleep disruption have been shown in various stages of abuse and recovery. Insomnia is the most well documented predictor of substance use relapse. Treatment specifically targeting chronic insomnia is essential for improved clinical outcomes. Although, chronic insomnia is a well-established, modifiable risk factor, to our knowledge, there are no interdisciplinary residential treatment programs that specifically treat chronic insomnia during acute SUDs treatment. We propose that improved treatment of insomnia as part of a comprehensive reinforcement-based outpatient treatment program will provide an efficient and cost effective opportunity to improve standard outpatient SUD. Converging evidence suggests that prophylactic CBT-I during SUD treatment may have short and long-term efficacy for sleep, and improve attrition. In the proposed study, patients with co-morbid SUDs and insomnia will engage in an 8-week group CBT-I (gCBT-I) program in addition to receiving treatment as usual for SUDs. This study may provide new hope to effectively treat insomnia in SUD and lead to a new standardization of outpatient care. We hypothesize that a CBT-I intervention can be implemented as part of an evidence-based SUD treatment program within a residential facility.

DETAILED DESCRIPTION:
Substance use disorders (SUDs) are a leading cause of global disease burden with significant epidemiological and economic consequences. Sleep disturbances (i.e., difficulty initiating or maintaining sleep) are nearly ubiquitous in individuals with SUDs and may arise from direct effects of the substance or from withdrawal of the substance. Sleep disturbances are reported in up to 70% of individuals entering both detoxification and early recovery programs and may persist for months to years during abstinence. Objective and subjective measures of sleep disturbances are among the best predictors of relapse. Treatment of insomnia (i.e., difficulty initiating or maintaining sleep, with significant daytime impairment) during early recovery may improve relapse rates. Insomnia is a modifiable risk factor and responds to psychological interventions. Given the abuse potential of many medications utilized for sleep disturbances and the likelihood of drug-drug interactions over the course of detoxification, a non-pharmacological approach to insomnia remains promising. To date, few studies have evaluated non-pharmacological approaches to insomnia during early substance abuse recovery. One study has evidenced improved self-reported sleep quality in men who were assigned to 2 weeks of daily progressive muscle relaxation training. Robust evidence indicates that cognitive behavioral therapy for insomnia (CBT-I) is effective, and in fact is first line treatment for primary insomnia. A preponderance of randomized controlled trials of CBT-I in co-morbid populations suggests it is efficacious to address insomnia in context of ongoing medical and psychiatric illnesses. Despite the possibility that treating insomnia may improve relapse and attrition rates, and evidence that CBT-I is efficacious in improving sleep, there is a dearth of empirical data regarding the prophylactic benefit of initiating CBT-I as part of acute abstinence treatment. This study aims to test the feasibility of implementing a non-pharmacological insomnia intervention for individuals at the Cornerstone clinic at the Helping Up Mission, a residential SUD residential recovery program for men in Baltimore, MD. Participants will be recruited from the Cornerstone clinic, an accredited behavioral health clinic directed by Johns Hopkins faculty and staff, which provides evidence-based SUD treatment to residents of the Helping Up Mission. CBT-I will be incorporated into the outpatient reinforcement-based SUD treatment. The investigators hypothesize that implementation of CBT-I during early SUD recovery is feasible and will lead to improved sleep parameters and improved clinical outcomes compared with those receiving treatment as usual (TAU). The investigators propose a proof of concept study which would first demonstrate feasibility of administering CBT-I for individuals residing in a men's homeless shelter, and will further evaluate the short- and long-term efficacy of CBT for insomnia in individuals with SUDs. This investigation will provide important and novel information regarding potential psychological interventions that may be incorporated into evidence-based SUD treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males > 18 years of age
* Active substance use disorder of any type
* Enrolled in the Cornerstone at Helping Up Mission clinic for less than 3 weeks
* ISI > 8
* Report either latency to sleep onset > 30 minutes or > 2 awakenings/night or > 15 min duration or wake after sleep onset (WASO) time > 30 minutes
* Insomnia symptom frequency self-reported as > 3 night/week for > 1 month

Exclusion Criteria:

* Self-report of Bipolar Disorder
* Self-report of Epilepsy or seizure disorder
* Suicidal ideation
* Acute Alcohol Withdrawal requiring medical attention

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Improvement in sleep. | Up to 6-month follow-up period.
  Participants in both study arms will record subjective sleep measures via self-report sleep diary. They will also complete the Insomnia Severity Index (ISI)) at both pre-and post-treatment and over 6-month follow-up period.

SECONDARY OUTCOMES:
Attrition in a substance abuse treatment program. | Up to 3-month follow-up period
  Attrition rates for the SUDs treatment program will be compared between the CBT-I and the treatment as usual group at 3-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Traci Speed, MD/PHD, Principal Investigator — Johns Hopkins University
Locations (1):
- Cornerstone at Helping Up Mission Clinic, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Speed TJ, Hanks L, Turner G, Gurule E, Kearson A, Buenaver L, Smith MT, Antoine D. A comparison of cognitive behavioral therapy for insomnia to standard of care in an outpatient substance use disorder clinic embedded within a therapeutic community: a RE-AIM framework evaluation. Trials. 2022 Nov 28;23(1):965. doi: 10.1186/s13063-022-06885-7. PMID 36443869